CLINICAL TRIAL: NCT06616376
Title: The Affect Of An Anti-Embolism Stocking Protocol On The Development Of Early Venous Thromboembolia In Patients With Knee Artroplasty
Brief Title: The Affect Of An Anti-Embolism Stocking Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ismail Furkan Basıbuyuk, specialist nurse, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CukurovaUBasibüyükErden
Record Dates: First submitted 2022-11-16; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Venous Thromboembolism
Keywords: Anti-embolism Stockings; Knee Arthroplasty; Nonpharmacological Method; Orthopedic Nursing; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: The study was conducted as a randomized controlled single-blind intervention study to determine the effect of the AES use protocol on the development of early VTE in patients undergoing knee arthroplasty.
Who Masked: Participant
Masking Description: To prevent patients undergoing TKA surgery from being affected by one another, the patients were hospitalized in separate rooms, and the orthopedic clinic team was made aware of the situation. The patients in the control group were told not to remove their socks until the sutures were removed after the operation, whereas the patients in the experimental group were told to remove their socks on the 10th day after the operation, so the patients had no idea which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): AES was redressed within the 21st day after the operation
  Interventions: Other: Anti-Embolism Stocking
- Control Group (No Intervention): The AES was dressed within the 10st day after the operation remained in the patient until the sutures

INTERVENTIONS:
Other: Anti-Embolism Stocking — To prevent patients undergoing TKA surgery from being affected by one another, the patients were hospitalized in separate rooms, and the orthopedic clinic team was made aware of the situation. The patients in the control group were told not to remove their socks until the sutures were removed after the operation, whereas the patients in the experimental group were told to remove their socks on the 10th day after the operation, so the patients had no idea which group they were in.
  Arms: Experimental Group

SUMMARY:
This study was conducted to determine the effect of anti-embolism stocking (AES) use protocol affected the development of early venous thromboembolism (VTE) in patients undergoing total knee arthroplasty (TKA).

The randomized controlled single-blind intervention study included 40 patients (Experimental Group: 20, Control Group: 20) who underwent TKA surgery in a university hospital's Orthopedics and Traumatology clinic between 2019 and 2021. While the experimental group received the AES protocol one day before the operation and continued until the 10 th day after the operation, the control group received AES on the 0 th day after the operation and remained in the patient until the 21st day after the operation. In the study, a "Data Collection Form" with DVT and PE signs and symptoms was used.

DETAILED DESCRIPTION:
The study was carried out at a university hospital's Orthopedics and Traumatology clinic. Knee arthroplasty surgery is performed on an average of 85 patients per year in the hospital with a bed capacity of 1200. The Orthopedics and Traumatology clinic has 36 beds and 9 nurses on staff.

In the clinic, LMWH is given to patients who will have knee arthroplasty 12 hours before the procedure. Following knee arthroplasty, an elastic bandage is placed over the dressing on the operated extremity, and AES is only applied to the intact extremity. AES is dressed on both extremities after the elastic bandage is removed. Foot movements begin on the first postoperative day, and patients are mobilized on the first or second postoperative day. Patients are admitted to the clinic for a period of 5-7 days. LMWH application, which began in the preoperative period, continues in the postoperative period for approximately 21 days (until the sutures are removed). The AES usage protocol is not implemented in the clinic, and no training is provided to patients regarding the use of AES by healthcare personnel. After TKA surgery, AES patients are dressed, and it is recommended that they wear them without removing them for 21 days (sutures are removed).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old,
* No harm in wearing AES,
* Patients who agreed to participate in the study.

Exclusion Criteria:

* Bilateral TKA used patients,
* Having excess leg edema, pulmonary edema, heart failure,
* Having leg ischemia,
* Having skin graft,
* An open wound in the area where AES will be applied,
* Having arterial and venous vessel disease,
* Having neuropathy,
* Having cellulite on the patient's leg to whom AES will be applied,
* Having an infection such as fasciitis or panniculitis,
* Those who declare that they will not use AES for ten days in accordance with the recommendations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Distribution of Descriptive Characteristics and Surgical Information of the Patients | Three weeks
  The mean age of the experimental group was 68.6±7.1 years (range: 51-81 years) and the mean age of the control group was 68.5±8.8 years (range: 57-89 years). There was chronic disease in 90% of the experimental group, and the rate of chronic disease in the control group was 60%. Mobility status of the experimental group 1 day before the surgery; 65% (n:13) were independent, 15% (n:3) self-supported and 20% (n:4) needed help. Mobility status of the control group 1 day before the surgery; 60% (n:11) were independent, 40% (n:8) self-supported, and 5% (n:1) needed help. Mobility status of the experimental group after surgery; 10% (n:2) were independent, 90% (n:18) were self-sufficient. Mobility status in the control group; 20% (n:4) were independent, 75% (n:15) were self-sufficient and 5% (n:1) needed help. All patients in the experimental and control groups used low molecular weight heparin or anticoagulants before surgery.
VTE Evaluation Form | Three weeks
  It consists of 19 questions covering symptoms of VTE, DVT and PE.

SECONDARY OUTCOMES:
The Use of Anti Embolism Stocking Protocol | Two weeks
  It Consısts Of 11 Questıons About The Use Of Antı-Embolısm Socks

CONTACTS AND LOCATIONS:
Overall Officials: Sevilay ERDEN, Assoc.Prof., Study Chair — Ç.Ü Faculty of Health Sciences Department of Surgical Nursing
Locations (1):
- Cukuruvo University, Adana, Sarıcam/Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-10-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT06616376/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT06616376/SAP_001.pdf